CLINICAL TRIAL: NCT04656496
Title: NOURISH-T+: A Randomized Control Trial Targeting Parents in Promoting Healthy Eating and Exercise Behaviors in Pediatric Cancer Survivors With Overweight/Obesity
Brief Title: NOURISH-T+: Promoting Healthy Eating and Exercise Behaviors
Acronym: NOURISH-T+
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: STUDY000244; R01CA240319 (NIH)
Record Dates: First submitted 2020-11-12; First posted 2020-12-07 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Obesity, Childhood; Cancer; Survivorship
MeSH Terms: conditions — Pediatric Obesity; Neoplasms

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NOURISH-T+ (Experimental): NOURISH-T+ targets parents as agents of change by providing intensive parent skills training emphasizing role modeling of positive health behaviors to foster the development of healthy eating and physical activity in pediatric cancer survivors. The NOURISH-T+ group will have 6 weekly, 1-1.5 hour, manualized sessions delivered using video-conferencing. There will be 2 additional brief sessions where the child will participate along with their parent to promote child engagement. Additionally, there will be one session with a pediatric oncology dietician based out of Nicklaus Children's Hospital who will discuss personalized nutritional strategies. Brief booster sessions at 2-, 4-, 8-, and 10- months will maximize retention and follow-up participation. NOURISH-T+ content is theory-based, manualized, and builds upon strengths of our prior work with NOURISH-T (our pilot) and NOURISH (our work with otherwise healthy overweight and obese children).
  Interventions: Behavioral: NOURISH-T+
- EUC - Brief NOURISH-T+ (Active Comparator): The EUC condition (Brief NOURISH-T+) engages parents in one information session moderated by a USF-based interventionist using videoconferencing. Session content is taken from the publicly available We Can! Manual. Parents in this group will receive nationally available web-based brochures on pediatric overweight/obesity on two occasions during the 6 weeks that NOURISH-T+ families participate in the study. Check-ins will take place at 2-, 4-, 8-, and 10- months post-intervention.
  Interventions: Behavioral: Brief NOURISH-T+

INTERVENTIONS:
Behavioral: NOURISH-T+ — NOURISH-T+ (Nourishing Our Understanding of Role Modeling to Improve Support and Healthy - Transitions) is a 6 session, psychoeducational program designed to teach parents of childhood cancer survivors with overweight/obesity knowledge and skills to improve the health and lifestyle behaviors for their child and for themselves.
  Arms: NOURISH-T+
Behavioral: Brief NOURISH-T+ — Enhanced Usual Care (or Brief NOURISH-T+) is an abbreviated version of the full NOURISH-T+ intervention in which parents are engaged in a one-time information session to also learn knowledge and skills to improve the health and lifestyle behaviors for their child and for themselves.
  Arms: EUC - Brief NOURISH-T+

SUMMARY:
Pediatric cancer survivors are at an increased risk of excessive weight gain and reduced exercise behaviors with the potential for this risk to worsen over time. With over 80% of pediatric cancer patients living to adulthood, many pediatric cancer survivors experience long-term health consequences such as heart disease - the leading cause of death in this population.

The purpose of this clinical research study is to teach parents/caregivers skills that will help prevent and reduce the problems of obesity in childhood cancer survivors. In this study, parents have the opportunity to participate in one of two web-based groups in which parents in either group will learn valuable information to improve the health of their child and of themselves.

DETAILED DESCRIPTION:
This project employs a cluster randomized, controlled, repeated measures trial study design, with parent-child dyads assigned to an evidence-informed manualized, social-cognitive parent intervention (NOURISH-T+) or to a comparison group (Enhanced Usual Care group - Brief NOURISH-T+). NOURISH-T+ stands for Nourishing Our Understanding of Role modeling to Improve Support and Health for Healthy Transitions.

Parents of pediatric cancer survivors (ages 5-14 years) with overweight and obesity, and off treatment for at least 6 months will be recruited across multiple pediatric oncology clinic sites. The University of South Florida (USF) serves as the coordinating data management and centralized research and intervention team and will also recruit eligible participants from its pediatric oncology clinic.

NOURISH-T+ targets parents as agents of change by providing intensive parent skills training emphasizing role modeling of positive health behaviors to foster the development of healthy eating and physical activity in pediatric cancer survivors. The NOURISH-T+ group will have 6 weekly, 1-1.5 hour, manualized sessions delivered using video-conferencing. There will be 2 additional brief sessions where the child will participate along with their parent to promote child engagement. Additionally, there will be one session with a pediatric oncology dietician based out of Nicklaus Children's Hospital who will discuss personalized nutritional strategies. Brief booster sessions at 2-, 4-, 8-, and 10- months will maximize retention and follow-up participation. NOURISH-T+ content is theory-based, manualized, and builds upon strengths of our prior work with NOURISH-T (our pilot) and NOURISH (our work with otherwise healthy overweight and obese children).

Parents randomized to Brief NOURISH-T+ will participate in one information session moderated by a USF-based interventionist using videoconferencing. Session content is taken from the publicly available We Can! Manual. Parents in this group will receive nationally available web-based brochures on pediatric overweight/obesity on two occasions during the 6 weeks that NOURISH-T+ families participate in the study. Check-ins will take place at 2-, 4-, 8-, and 10- months post-intervention.

Outcome measures will be completed at baseline, 3-, 6-, and 12-months post-intervention.

ELIGIBILITY:
Inclusion Criteria:

Eligible Pediatric Cancer Survivors must be:

1. 5-14 years of age at enrollment;
2. Off active treatment for at least 6 months;
3. At or above the 85th BMI %ile;
4. Able to complete assessments with the help of clinic staff and the USF research team;
5. Residing with the participating parent;
6. Able to engage in PA tailored to current medical status;
7. NOT taking medications that affect body weight (e.g., steroids) within 6 months of enrollment, and
8. In remission -- PCS who experience a relapse of cancer during the intervention will be excused from further involvement.
9. Must be English- or Spanish-speaking

Participating Parents must:

* Be either biological or adoptive and/or step mothers or fathers and must be permanent legal guardians of the PCS
* Be at least 18 years old
* Identifies as the main meal preparer at home
* Must be English- or Spanish-speaking

Exclusion Criteria:

* Parents are ineligible if they are non-ambulatory and/or do not reside at least 50% of the time with their participating child.
* Female parents who are currently pregnant will be excluded from the study.
* Children are ineligible to participate if they are non-ambulatory. In addition, children who are wards of the state will be excluded from the study.

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 520 (Estimated)
Dates: Start 2020-12-08 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in Child BMI z-score | baseline to 6 months
  Height and weight will be measured to obtain BMI z-score for gender and age.
Change in Child BMI z-score | baseline to 12 months
  Height and weight will be measured to obtain BMI z-score for gender and age.

SECONDARY OUTCOMES:
Change in Child Physical Activity Behaviors | baseline to 6 months
  Waist-worn accelerometers will be worn for one week to calculate average daily step count over one week. Accelerometers objectively measure daily PA, including average steps per day, time spent in moderate-vigorous activity, and sedentary time.
Change in Child Physical Activity Behaviors | baseline to 12 months
  Waist-worn accelerometers will be worn for one week to calculate average daily step count over one week. Accelerometers objectively measure daily PA, including average steps per day, time spent in moderate-vigorous activity, and sedentary time.
Change in Child Eating Behaviors | baseline to 6 months
  Dietary Recall Automated Self-administered 24-Hour Dietary Recall-2020(ASA24). ASA24 is a highly reliable, computer assisted 24-hour dietary recall interview with animated guides and audio and visual cues to instruct participants and enhance use in low-literacy populations.
Change in Child Eating Behaviors | baseline to 12 months
  Dietary Recall Automated Self-administered 24-Hour Dietary Recall-2020(ASA24). ASA24 is a highly reliable, computer assisted 24-hour dietary recall interview with animated guides and audio and visual cues to instruct participants and enhance use in low-literacy populations.
Change in Parent BMI | baseline to 6 months
  Height and weight will be measured and used to calculate continuous adult BMI score.
Change in Parent BMI | baseline to 12 months
  Height and weight will be measured and used to calculate continuous adult BMI score.

CONTACTS AND LOCATIONS:
Overall Officials: Marilyn Stern, PhD, Principal Investigator — University of South Florida
Locations (10):
- United States (10):
  - Children's National Hospital, Washington D.C., District of Columbia
  - University of Florida Health System, Gainesville, Florida
  - University of Miami Health System, Miami, Florida
  - Nicklaus Children's Hospital, Miami, Florida
  - USF Pediatrics, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Johns Hopkins Medicine, Baltimore, Maryland
  - Washington University School of Medicine, St Louis, Missouri
  - Hackensack Meridian Health, Hackensack, New Jersey
  - Virginia Commonwealth University, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ruble K, Davis CL, Han HR. Endothelial health in childhood acute lymphoid leukemia survivors: pilot evaluation with peripheral artery tonometry. J Pediatr Hematol Oncol. 2015 Mar;37(2):117-20. doi: 10.1097/MPH.0000000000000122. PMID 24577544
- [Background] Ruble K, Scarvalone S, Gallicchio L, Davis C, Wells D. Group Physical Activity Intervention for Childhood Cancer Survivors: A Pilot Study. J Phys Act Health. 2016 Mar;13(3):352-9. doi: 10.1123/jpah.2015-0050. Epub 2015 Aug 13. PMID 26284383
- [Background] Nathan PC, Ford JS, Henderson TO, Hudson MM, Emmons KM, Casillas JN, Lown EA, Ness KK, Oeffinger KC. Health behaviors, medical care, and interventions to promote healthy living in the Childhood Cancer Survivor Study cohort. J Clin Oncol. 2009 May 10;27(14):2363-73. doi: 10.1200/JCO.2008.21.1441. Epub 2009 Mar 2. PMID 19255308
- [Background] Stull VB, Snyder DC, Demark-Wahnefried W. Lifestyle interventions in cancer survivors: designing programs that meet the needs of this vulnerable and growing population. J Nutr. 2007 Jan;137(1 Suppl):243S-248S. doi: 10.1093/jn/137.1.243S. PMID 17182834
- [Background] Reilly JJ, Blacklock CJ, Dale E, Donaldson M, Gibson BE. Resting metabolic rate and obesity in childhood acute lymphoblastic leukaemia. Int J Obes Relat Metab Disord. 1996 Dec;20(12):1130-2. PMID 8968860
- [Background] Greving DM, Santacroce SJ. Cardiovascular late effects. J Pediatr Oncol Nurs. 2005 Jan-Feb;22(1):38-47. doi: 10.1177/1043454204272531. PMID 15574725
- [Background] Oeffinger KC, Mertens AC, Sklar CA, Yasui Y, Fears T, Stovall M, Vik TA, Inskip PD, Robison LL; Childhood Cancer Survivor Study. Obesity in adult survivors of childhood acute lymphoblastic leukemia: a report from the Childhood Cancer Survivor Study. J Clin Oncol. 2003 Apr 1;21(7):1359-65. doi: 10.1200/JCO.2003.06.131. PMID 12663727
- [Background] Chow EJ, Pihoker C, Hunt K, Wilkinson K, Friedman DL. Obesity and hypertension among children after treatment for acute lymphoblastic leukemia. Cancer. 2007 Nov 15;110(10):2313-20. doi: 10.1002/cncr.23050. PMID 17896787
- [Background] Mayer EI, Reuter M, Dopfer RE, Ranke MB. Energy expenditure, energy intake and prevalence of obesity after therapy for acute lymphoblastic leukemia during childhood. Horm Res. 2000;53(4):193-9. doi: 10.1159/000023566. PMID 11044803
- [Background] Warner JT. Body composition, exercise and energy expenditure in survivors of acute lymphoblastic leukaemia. Pediatr Blood Cancer. 2008 Feb;50(2 Suppl):456-61; discussion 468. doi: 10.1002/pbc.21411. PMID 18064643
- [Background] Ness KK, Leisenring WM, Huang S, Hudson MM, Gurney JG, Whelan K, Hobbie WL, Armstrong GT, Robison LL, Oeffinger KC. Predictors of inactive lifestyle among adult survivors of childhood cancer: a report from the Childhood Cancer Survivor Study. Cancer. 2009 May 1;115(9):1984-94. doi: 10.1002/cncr.24209. PMID 19224548
- [Background] Zhang FF, Rodday AM, Kelly MJ, Must A, MacPherson C, Roberts SB, Saltzman E, Parsons SK. Predictors of being overweight or obese in survivors of pediatric acute lymphoblastic leukemia (ALL). Pediatr Blood Cancer. 2014 Jul;61(7):1263-9. doi: 10.1002/pbc.24960. Epub 2014 Jan 30. PMID 24482072
- [Background] Cox CL, Montgomery M, Oeffinger KC, Leisenring W, Zeltzer L, Whitton JA, Mertens AC, Hudson MM, Robison LL. Promoting physical activity in childhood cancer survivors: results from the Childhood Cancer Survivor Study. Cancer. 2009 Feb 1;115(3):642-54. doi: 10.1002/cncr.24043. PMID 19117349
- [Background] Clarke SA, Eiser C. Health behaviours in childhood cancer survivors: a systematic review. Eur J Cancer. 2007 Jun;43(9):1373-84. doi: 10.1016/j.ejca.2007.03.002. Epub 2007 Apr 24. PMID 17459696
- [Background] Armstrong GT, Oeffinger KC, Chen Y, Kawashima T, Yasui Y, Leisenring W, Stovall M, Chow EJ, Sklar CA, Mulrooney DA, Mertens AC, Border W, Durand JB, Robison LL, Meacham LR. Modifiable risk factors and major cardiac events among adult survivors of childhood cancer. J Clin Oncol. 2013 Oct 10;31(29):3673-80. doi: 10.1200/JCO.2013.49.3205. Epub 2013 Sep 3. PMID 24002505
- [Background] Oeffinger KC, Mertens AC, Sklar CA, Kawashima T, Hudson MM, Meadows AT, Friedman DL, Marina N, Hobbie W, Kadan-Lottick NS, Schwartz CL, Leisenring W, Robison LL; Childhood Cancer Survivor Study. Chronic health conditions in adult survivors of childhood cancer. N Engl J Med. 2006 Oct 12;355(15):1572-82. doi: 10.1056/NEJMsa060185. PMID 17035650
- [Background] Hudson MM, Mertens AC, Yasui Y, Hobbie W, Chen H, Gurney JG, Yeazel M, Recklitis CJ, Marina N, Robison LR, Oeffinger KC; Childhood Cancer Survivor Study Investigators. Health status of adult long-term survivors of childhood cancer: a report from the Childhood Cancer Survivor Study. JAMA. 2003 Sep 24;290(12):1583-92. doi: 10.1001/jama.290.12.1583. PMID 14506117
- [Background] Eiser C. Beyond survival: quality of life and follow-up after childhood cancer. J Pediatr Psychol. 2007 Oct;32(9):1140-50. doi: 10.1093/jpepsy/jsm052. Epub 2007 Jul 20. PMID 17644535
- [Background] Green D, Wallace H. Late effects of Childhood Cancer. CRC Press; 2003.
- [Background] Smith AW, Baum A, Wing RR. Stress and weight gain in parents of cancer patients. Int J Obes (Lond). 2005 Feb;29(2):244-50. doi: 10.1038/sj.ijo.0802835. PMID 15654361
- [Background] Lipshultz SE, Adams MJ, Colan SD, Constine LS, Herman EH, Hsu DT, Hudson MM, Kremer LC, Landy DC, Miller TL, Oeffinger KC, Rosenthal DN, Sable CA, Sallan SE, Singh GK, Steinberger J, Cochran TR, Wilkinson JD; American Heart Association Congenital Heart Defects Committee of the Council on Cardiovascular Disease in the Young, Council on Basic Cardiovascular Sciences, Council on Cardiovascular and Stroke Nursing, Council on Cardiovascular Radiolo. Long-term cardiovascular toxicity in children, adolescents, and young adults who receive cancer therapy: pathophysiology, course, monitoring, management, prevention, and research directions: a scientific statement from the American Heart Association. Circulation. 2013 Oct 22;128(17):1927-95. doi: 10.1161/CIR.0b013e3182a88099. Epub 2013 Sep 30. No abstract available. PMID 24081971
- [Background] Stolley MR, Sharp LK, Tangney CC, Schiffer LA, Arroyo C, Kim Y, Campbell RT, Schmidt ML, Breen K, Kinahan KE, Dilley KJ, Henderson TO, Korenblit AD, Seligman K. Health behaviors of minority childhood cancer survivors. Cancer. 2015 May 15;121(10):1671-80. doi: 10.1002/cncr.29202. Epub 2015 Jan 6. PMID 25564774
- [Background] Sklar CA, Mertens AC, Walter A, Mitchell D, Nesbit ME, O'Leary M, Hutchinson R, Meadows AT, Robison LL. Changes in body mass index and prevalence of overweight in survivors of childhood acute lymphoblastic leukemia: role of cranial irradiation. Med Pediatr Oncol. 2000 Aug;35(2):91-5. doi: 10.1002/1096-911x(200008)35:23.0.co;2-g. PMID 10918229
- [Background] Stern M, Bachar E, Ronen Ackerman E, Rancourt D, Bonne O, Weintraub M. Weight Trajectories of Israeli Pediatric Cancer Survivors. J Pediatr Psychol. 2017 Jun 1;42(5):588-597. doi: 10.1093/jpepsy/jsw102. PMID 28130395
- [Background] Ogden CL, Carroll MD, Kit BK, Flegal KM. Prevalence of obesity and trends in body mass index among US children and adolescents, 1999-2010. JAMA. 2012 Feb 1;307(5):483-90. doi: 10.1001/jama.2012.40. Epub 2012 Jan 17. PMID 22253364
- [Background] Zhang FF, Parsons SK. Obesity in Childhood Cancer Survivors: Call for Early Weight Management. Adv Nutr. 2015 Sep 15;6(5):611-9. doi: 10.3945/an.115.008946. Print 2015 Sep. PMID 26374183
- [Background] Moyer A, Knapp-Oliver SK, Sohl SJ, Schnieder S, Floyd AH. Lessons to be learned from 25 years of research investigating psychosocial interventions for cancer patients. Cancer J. 2009 Sep-Oct;15(5):345-51. doi: 10.1097/PPO.0b013e3181bf51fb. PMID 19826351
- [Background] van Brussel M, Takken T, Lucia A, van der Net J, Helders PJ. Is physical fitness decreased in survivors of childhood leukemia? A systematic review. Leukemia. 2005 Jan;19(1):13-7. doi: 10.1038/sj.leu.2403547. PMID 15526028
- [Background] Warner JT, Bell W, Webb DK, Gregory JW. Daily energy expenditure and physical activity in survivors of childhood malignancy. Pediatr Res. 1998 May;43(5):607-13. doi: 10.1203/00006450-199805000-00008. PMID 9585006
- [Background] Mazzeo SE, Kelly NR, Stern M, Gow RW, Serdar K, Evans RK, Jones RM, Bulik CM. Nourishing Our Understanding of Role Modeling to Improve Support and Health (NOURISH): design and methods. Contemp Clin Trials. 2012 May;33(3):515-22. doi: 10.1016/j.cct.2012.01.003. Epub 2012 Jan 18. PMID 22273843
- [Background] Mackinnon DP. Integrating Mediators and Moderators in Research Design. Res Soc Work Pract. 2011 Nov;21(6):675-681. doi: 10.1177/1049731511414148. Epub 2011 Jul 13. PMID 22675239
- [Background] Lydecker JA, Simpson C, Kwitowski M, Gow RW, Stern M, Bulik CM, Mazzeo SE. Evaluation of Parent-Reported Feeding Practices in a Racially Diverse, Treatment-Seeking Child Overweight/Obesity Sample. Child Health Care. 2017;46(3):265-281. doi: 10.1080/02739615.2016.1163489. Epub 2016 Mar 17. PMID 28959085
- [Background] Stern, M., Mazzeo, S.E., Porter, J. et al. Self-Esteem, Teasing and Quality of Life: African American Adolescent Girls Participating in a Family-Based Pediatric Overweight Intervention. J Clin Psychol Med Settings 13, 217 (2006). https://doi.org/10.1007/s10880-006-9029-4
- [Background] Stern M, Ewing L, Davila E, Thompson AL, Hale G, Mazzeo S. Design and rationale for NOURISH-T: a randomized control trial targeting parents of overweight children off cancer treatment. Contemp Clin Trials. 2015 Mar;41:227-37. doi: 10.1016/j.cct.2014.12.018. Epub 2015 Jan 2. PMID 25559916
- [Background] Bean MK, Wilson DB, Thornton LM, Kelly N, Mazzeo SE. Dietary intake in a randomized-controlled pilot of NOURISH: a parent intervention for overweight children. Prev Med. 2012 Sep;55(3):224-7. doi: 10.1016/j.ypmed.2012.06.016. Epub 2012 Jun 24. PMID 22735041
- [Background] Raber M, Swartz MC, Santa Maria D, O'Connor T, Baranowski T, Li R, Chandra J. Parental involvement in exercise and diet interventions for childhood cancer survivors: a systematic review. Pediatr Res. 2016 Sep;80(3):338-46. doi: 10.1038/pr.2016.84. Epub 2016 Apr 11. PMID 27064243
- [Background] Epstein LH, Valoski A, Wing RR, McCurley J. Ten-year outcomes of behavioral family-based treatment for childhood obesity. Health Psychol. 1994 Sep;13(5):373-83. doi: 10.1037//0278-6133.13.5.373. PMID 7805631
- [Background] Epstein LH, Valoski A, Wing RR, McCurley J. Ten-year follow-up of behavioral, family-based treatment for obese children. JAMA. 1990 Nov 21;264(19):2519-23. PMID 2232019
- [Background] Epstein LH, Wing RR, Koeske R, Andrasik F, Ossip DJ. Child and parent weight loss in family-based behavior modification programs. J Consult Clin Psychol. 1981 Oct;49(5):674-85. doi: 10.1037//0022-006x.49.5.674. No abstract available. PMID 7287977
- [Background] Epstein LH, Wing RR, Koeske R, Valoski A. Long-term effects of family-based treatment of childhood obesity. J Consult Clin Psychol. 1987 Feb;55(1):91-5. doi: 10.1037//0022-006x.55.1.91. No abstract available. PMID 3106445
- [Background] Golan M, Crow S. Parents are key players in the prevention and treatment of weight-related problems. Nutr Rev. 2004 Jan;62(1):39-50. doi: 10.1111/j.1753-4887.2004.tb00005.x. PMID 14995056
- [Background] Golan M. Parents as agents of change in childhood obesity--from research to practice. Int J Pediatr Obes. 2006;1(2):66-76. doi: 10.1080/17477160600644272. PMID 17907317
- [Background] Kitzmann KM, Dalton WT 3rd, Stanley CM, Beech BM, Reeves TP, Buscemi J, Egli CJ, Gamble HL, Midgett EL. Lifestyle interventions for youth who are overweight: a meta-analytic review. Health Psychol. 2010 Jan;29(1):91-101. doi: 10.1037/a0017437. PMID 20063940
- [Background] Smith JD, Berkel C, Jordan N, Atkins DC, Narayanan SS, Gallo C, Grimm KJ, Dishion TJ, Mauricio AM, Rudo-Stern J, Meachum MK, Winslow E, Bruening MM. An individually tailored family-centered intervention for pediatric obesity in primary care: study protocol of a randomized type II hybrid effectiveness-implementation trial (Raising Healthy Children study). Implement Sci. 2018 Jan 15;13(1):11. doi: 10.1186/s13012-017-0697-2. PMID 29334983
- [Background] Stern M, Bleck J, Ewing LJ, Davila E, Lynn C, Hale G, Mazzeo S. NOURISH-T: Targeting caregivers to improve health behaviors in pediatric cancer survivors with obesity. Pediatr Blood Cancer. 2018 May;65(5):e26941. doi: 10.1002/pbc.26941. Epub 2018 Jan 19. PMID 29350459
- [Background] Stern, M., Lamanna, J., Russell, C., Ewing, L., Thompson, A., Trapp, S., Bitsko, M., & Mazzeo, S. (2013). Adaptation of an obesity intervention program for pediatric cancer survivors (NOURISH-T). Clinical Practice in Pediatric Psychology, 1(3), 264-275. https://doi.org/10.1037/cpp0000023
- [Background] Mazzeo S, Gow R, Stern M, Gerke C. Developing an intervention for parents of overweight children. International Journal of Child and Adolescent Health. 2008;1(4):355-363.
- [Derived] Brown NI, Sauls R, Almendares M, Gray HL, Stern M. Factors impacting physical activity among post-treatment pediatric cancer survivors with overweight and obesity. Eur J Pediatr. 2024 Jul;183(7):3129-3136. doi: 10.1007/s00431-024-05584-6. Epub 2024 Apr 26. PMID 38668797
- [Derived] Buro AW, Gray HL, Ruble K, Soca Lozano S, Sauls R, Albizu-Jacob A, Crowder SL, Mazzeo SE, Stern M. Challenges and adaptations for a cluster-randomized control trial targeting parents of pediatric cancer survivors with obesity during the COVID-19 pandemic. Transl Behav Med. 2023 Feb 28;13(2):98-103. doi: 10.1093/tbm/ibac084. PMID 36327379
- [Derived] Stern M, Gray HL, Ruble K, Soca Lozano S, Albizu-Jacob A, Williams JM, Godder K, Fuemmeler B, Mazzeo S. A cluster-randomized control trial targeting parents of pediatric cancer survivors with obesity: Rationale and study protocol of NOURISH-T. Contemp Clin Trials. 2021 Mar;102:106296. doi: 10.1016/j.cct.2021.106296. Epub 2021 Jan 27. PMID 33515782